CLINICAL TRIAL: NCT04675944
Title: An Open-Label, Three Period, Fixed Sequence Study to Assess the Effect of a Single Dose of BIA 5 1058 200 mg on the Steady State Pharmacokinetics of Treprostinil in Healthy Subjects Under Fed Conditions
Brief Title: Effect of BIA 5-1058 on the Steady State Pharmacokinetics of Treprostinil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BIA-51058-106; 2017-000245-43 (EudraCT Number)
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — zamicastat; treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BIA 5-1058 / treprostinil (Experimental): Three treatment periods separated by a washout period of at least 10 days
  Interventions: Drug: BIA 5-1058; Drug: treprostinil

INTERVENTIONS:
Drug: BIA 5-1058 — 200 mg (2 x 100 mg tablets), oral route
  Other Names: Zamicastat
Drug: treprostinil — 1 mg (1 extended-release tablet), oral route
  Other Names: Orenitram

SUMMARY:
The purpose of this study is to assess the effect of BIA 5-1058 200 mg on the pharmacokinetic (PK) of treprostinil

DETAILED DESCRIPTION:
This study was an open-label, three period, fixed sequence study in healthy male and female subjects performed at a single study center.

The study comprised:

* Screening during Days -28 to -2 (both inclusive).
* Three treatment periods separated by a washout period of at least 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. Provided a signed and dated informed consent before any study specific procedures were conducted.
2. Male and female subjects aged 18 to 45 years (both inclusive) at the Screening Visit.
3. Healthy as determined by the Principal Investigator based on medical history, physical examination, clinical laboratory test results, vital signs and digital 12 lead electrocardiogram (ECG). If a vital sign or ECG assessment was outside of the reference range at the Screening Visit or baseline, the assessment could have been repeated once as soon as possible and in any cases before enrolment to rule out any error.
4. Non-smoker or ex-smoker for at least 3 months prior to the Screening Visit.
5. Body mass index (BMI) between 18.5 and 29.9 kg/m2 (both inclusive) at the Screening Visit and on admission to each treatment period.
6. Negative test results for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (anti HBc), immunoglobulin M (IgM) anti-HBc, hepatitis C virus antibody (anti HCV) and human immunodeficiency virus (HIV) (Types 1 and 2) antibodies at the Screening Visit.
7. Negative screen for alcohol and drugs of abuse at the Screening Visit and on admission to each treatment period.
8. Subject had to be willing and able to be confined to the clinical unit and had to adhere to the study and lifestyle restrictions.
9. Contraception requirements:

Male subjects had to use together with his female partner/spouse a highly effective contraception form of birth control in combination with a barrier method throughout the clinical study period and agreed not to father a child or to donate sperm starting at the Screening Visit and throughout the clinical study.

Female subjects had to either be of non childbearing potential or had to use highly effective methods of contraception from at least 3 months before the Screening Visit and throughout the clinical study in combination with a barrier method.

Exclusion Criteria:

Inclusion Criteria:

Subjects who met the following criteria were considered eligible to participate/continue in the study:

1. Provided a signed and dated informed consent before any study specific procedures were conducted.
2. Male and female subjects aged 18 to 45 years (both inclusive) at the Screening Visit.
3. Healthy as determined by the Principal Investigator based on medical history, physical examination, clinical laboratory test results, vital signs and digital 12 lead electrocardiogram (ECG). If a vital sign or ECG assessment was outside of the reference range at the Screening Visit or baseline, the assessment could have been repeated once as soon as possible and in any cases before enrolment to rule out any error.
4. Non-smoker or ex-smoker for at least 3 months prior to the Screening Visit.
5. Body mass index (BMI) between 18.5 and 29.9 kg/m2 (both inclusive) at the Screening Visit and on admission to each treatment period.
6. Negative test results for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (anti HBc), immunoglobulin M (IgM) anti-HBc, hepatitis C virus antibody (anti HCV) and human immunodeficiency virus (HIV) (Types 1 and 2) antibodies at the Screening Visit.
7. Negative screen for alcohol and drugs of abuse at the Screening Visit and on admission to each treatment period.
8. Subject had to be willing and able to be confined to the clinical unit and had to adhere to the study and lifestyle restrictions.
9. Contraception requirements:

Male subjects had to use together with his female partner/spouse a highly effective contraception form of birth control in combination with a barrier method throughout the clinical study period and agreed not to father a child or to donate sperm starting at the Screening Visit and throughout the clinical study.

Female subjects had to either be of non childbearing potential or had to use highly effective methods of contraception from at least 3 months before the Screening Visit and throughout the clinical study in combination with a barrier method.

Exclusion Criteria:

Subjects that met any of the following criteria were not considered eligible to participate/continue in the study:

1. Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue disease or disorders within 5 years before the first investigational medicinal product (IMP) administration.
2. Documented coronary artery disease (any of prior myocardial infarction, positive stress test, positive nuclear perfusion study, prior coronary artery bypass graft [CABG] surgery or percutaneous coronary intervention, angiogram showing at least 75% stenosis in a major coronary artery), acute coronary syndrome or current symptoms of myocardial ischemia and angina.
3. Clinically relevant surgical history that involved the stomach and/or intestinal system, potentially affecting absorption of IMPs.
4. Any clinically relevant findings in the laboratory tests, particularly any abnormality in the coagulation tests or the liver function tests, as judged by the Principal Investigator, at the Screening Visit and on admission to each treatment period. If a laboratory assessment was outside of the reference range at the local laboratory at the Screening Visit or baseline, the assessment could have been repeated once as soon as possible and in any cases before enrolment to rule out laboratory error.
5. Subjects with alanine aminotransferase (ALT) > 1.0 x the upper limit of normal (ULN) and/or aspartate aminotransferase (AST) > 1.0 x ULN and/or total bilirubin > 1.0 x ULN (isolated bilirubin > 1.0 x ULN and ≤ 1.5 x ULN was acceptable if bilirubin was fractionated and direct bilirubin < 35%), as confirmed by subsequent repeat assessment, at the Screening Visit and on admission to each treatment period.
6. History of relevant atopy or drug hypersensitivity.
7. History of alcoholism or drug abuse.
8. History of drinking > 24 g (males) and > 12 g (females) of pure alcohol per day (10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) within 3 months before first admission to the clinical unit.
9. Use of alcohol within 72 hours before the Screening Visit and from 48 hours before dosing until completion of the Follow-up Visit.
10. Significant infection or known inflammatory process at the Screening Visit or upon admission to all Treatment Periods, as judged by the Principal Investigator.
11. Acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhea, heartburn) at the time of the Screening Visit or upon admission to all treatment periods.
12. Subjects with blood pressure (BP) measurements (mean of triplicate) outside the ranges, at the Screening Visit or admission to the first treatment period:

    * Systolic blood pressure (SBP) < 100 mmHg or > 140 mmHg
    * Diastolic blood pressure (DBP) < 60 mmHg or > 90 mmHg
13. Symptomatic orthostatic hypotension (drop of > 20 mmHg in SBP and/or > 10 mmHg in DBP when moving from supine to standing position), together with other symptoms, e.g., dizziness, at the Screening Visit or admission to the first treatment Period.
14. Abnormal fundoscopy.
15. Electrocardiogram (mean of triplicate) with corrected QT interval using the Fridericia's formula (QTcF) > 450 ms at the Screening Visit or admission to the first treatment period.
16. Having an estimated glomerular filtration rate (eGFR) < 90 mL/min, based on creatinine clearance calculation by the Cockcroft Gault formula and normalized to an average surface area of 1.73m2.
17. Previous use of BIA 5 1058.
18. Use of any investigational drug or participation in any clinical study within 60 days or 5 half life times, whichever was longer, before the first administration of IMP.
19. Having received IMP in more than 3 studies within 12 months before the Screening Visit.
20. Donated or received blood within 56 days before first administration of IMP.
21. Donated or received plasma within 30 days before first administration of IMP.
22. History of any significant bleeding within the last 56 days prior to first administration of IMP.
23. Vegetarians, vegans or other medical dietary restrictions.
24. Not able to communicate reliably with the Principal Investigator.
25. Unlikely to comply with the requirements of the study.
26. Use of over the counter (OTC) medications (including oral natural health products, vitamin, and herbal supplements) within 7 days before the first IMP administration until the Follow up Visit.

    * Use of prescription medications that could have affected the safety or other study assessments, in the Principal Investigator's opinion, within 14 days before the first IMP administration until the Follow-up Visit. By exception, acetaminophen/paracetamol -1000 mg/day was permitted.
    * CYP2B6, CYP2C8, CYP2D6, CYP3A4 (BIA 5-1058 metabolism) and CYP2C9, CYP2C8 (treprostinil metabolism): use of inhibitors taken within 7 days before the first IMP administration and inducers taken within 28 days before first IMP administration.
27. Any known allergy or contraindication to any of the IMPs or their content.
28. The subject was an employee or the close relative of an employee of the Sponsor or the Contract Research Organization (CRO) involved in the clinical study.
29. Vulnerable subjects, e.g., subjects kept in detention, protected adults under guardianship, trusteeship and soldiers or subjects committed to an institution by governmental or juridical order.

    If female:
30. Pregnant or breastfeeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration - Cmax | Pre-dose (Treatment Period 1, Day 1 and Treatment Period 3, Day 6) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours
  Primary Pharmacokinetic Parameters - BIA 5 1058
Area under the plasma concentration-time curve (AUC) from time zero to the last quantifiable concentration - AUC0-t | Pre-dose (Treatment Period 1, Day 1 and Treatment Period 3, Day 6) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours
  Primary Pharmacokinetic Parameters - BIA 5 1058
AUC from time zero extrapolated to infinity - AUC0-inf | Pre-dose (Treatment Period 1, Day 1 and Treatment Period 3, Day 6) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours
  Primary Pharmacokinetic Parameters - BIA 5 1058
Maximum observed plasma concentration at steady state - Cmax,ss | Pre-last dose (Treatment Period 2, Day 6 and Treatment Period 3, Day 6) and post-last dose at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours.
  Primary Pharmacokinetic Parameters - Treprostinil
AUC over the dosing interval at steady state - AUC0-τ,ss | Pre-last dose (Treatment Period 2, Day 6 and Treatment Period 3, Day 6) and post-last dose at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours.
  Primary Pharmacokinetic Parameters - Treprostinil

CONTACTS AND LOCATIONS:
Locations (1):
- PAREXEL International - Early Phase Clinical Unit, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided